CLINICAL TRIAL: NCT01657331
Title: A Phase I/II Clinical Trial of the Combination of Brentuximab Vedotin and Bendamustine in Patients With Relapsed or Refractory Hodgkin Lymphoma or Anaplastic Large Cell Lymphoma
Brief Title: Brentuximab Vedotin and Bendamustine for the Treatment of Hodgkin Lymphoma and Anaplastic Large Cell Lymphoma (ALCL)
Acronym: SGN+Benda
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAJ5050
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Hodgkin Lymphoma; Anaplastic Large Cell Lymphoma
Keywords: Hodgkin Lymphoma; Hodgkin Disease; Hodgkin's Disease; Anaplastic Large Cell Lymphoma; ALCL; SGN+Benda; Bendamustine; Brentuximab Vedotin
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic | interventions — Brentuximab Vedotin; Bendamustine Hydrochloride; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brentuximab Vedotin / Bendamustine (Experimental): Subjects with relapsed or refractory Hodgkin Lymphoma or Anaplastic Large Cell Lymphoma will receive Brentuximab Vedotin in combination with Bendamustine, and prophylactic Neulasta
  Interventions: Drug: Brentuximab Vedotin; Drug: Bendamustine; Drug: Neulasta

INTERVENTIONS:
Drug: Brentuximab Vedotin — Dose escalation in phase I of the study from 1.2-1.8 mg/kg, IV infusions over 30 minutes on day 1 of each 21-day cycle.
  Other Names: Adcetris; SGN35
Drug: Bendamustine — Dose escalation in phase I of the study from 60-100 mg/m2, IV infusion on days 1 and 2 of each 21-day cycle.
  Other Names: Treanda; Bendamustine HCl
Drug: Neulasta — (Non-experimental) Standard procedure prophylactic pegfilgrastim on day 3 of any subsequent cycle after cycle 1, or filgrastim for 5 to 10 days, per investigator's discretion.
  Other Names: pegfilgrastim

SUMMARY:
This is a phase 1/2 multicenter study to assess the safety and effectiveness of brentuximab vedotin and bendamustine, when given together, in patients with Hodgkin Lymphoma or Anaplastic Large Cell Lymphoma (ALCL) that has either returned or did not respond to initial treatment(s). Patients will be accrued at Columbia University Medical Center (CUMC) and at two subsites in Canada.

DETAILED DESCRIPTION:
Brentuximab vedotin will be administered as an outpatient IV infusion on day 1 of each 21-day cycle. Bendamustine will be given as an outpatient infusion on days 1 and 2 of a 21-day cycle. Patients may receive prophylactic pegfilgrastim on day 3 of each cycle, or filgrastim for 5 to 10 days, per investigator's discretion. Patients can receive a maximum of 6 cycles of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed relapsed or refractory HL or ALCL.
* Documented CD30+ expression from either original diagnosis or a tumor biopsy in the relapsed setting.
* For patients with HL, subjects are eligible after failure or having declined autologous stem cell transplant or at least two prior multi-agent chemotherapy regimens if they are not autologous stem cell transplant candidates. For patients with ALCL, subjects are eligible after failure of at least one prior multi-agent chemotherapy regimen and if they are not eligible for or have declined autologous stem cell transplant.
* Must have received first line chemotherapy. No upper limit for the number of prior therapies.
* Patients with prior autologous or allogeneic stem cell transplant are eligible as long as they meet all other criteria.
* Measurable or evaluable disease, as defined in 2008 Revised Response Criteria for Malignant Lymphoma(33)
* Age > or = 18 years
* ECOG performance status 0,1 or 2
* Patient's must have adequate organ and marrow function as defined below

  * Absolute neutrophil count > or = 1,000 (1.0 x 109/L)
  * Platelets > or = 50,000 (50 x 109/L)
  * Total Bilirubin < or = 1.5 x institutional limits unless documented Gilbert's syndrome (then < 2.5 x institutional upper limit)
  * AST (SGOT)/ALT (SGPT) < or = 2.0 x institutional upper limit of normal (unless known hepatic involvement then < 3.5 x institutional upper limit)
  * Creatinine within normal institutional limits OR creatinine clearance > or = 50mL/min for patients with creatinine levels above institutional normal
* If female of childbearing age, negative serum pregnancy test within 7 days prior to the first dose of brentuximab vedotin in this study
* Must be willing to use contraception during the study, and for 30 days following the last dose of study drug.
* Able to understand and to sign a written consent document

Exclusion Criteria:

* Prior treatment with brentuximab vedotin and bendamustine in combination. May have received prior therapy with brentuximab vedotin or bendamustine separately.
* Received either brentuximab vedotin or bendamustine within 3 months of receiving their first dose of protocol based therapy.
* If brentuximab vedotin or bendamustine was previously received, had disease progression during the first 3 cycles of either brentuximab vedotin or bendamustine.
* Systemic steroids that have not been stabilized to the equivalent of < 10 mg/day of prednisone 7 days prior to the initiation of the trial.
* ANY concurrent investigational agents.
* Exposure to chemotherapy, radiotherapy, biologics or investigational agents within 3 weeks prior enrollment in the study.
* Known cerebral or meningeal disease.
* Active concurrent malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix). If there is a history of prior malignancy the patients must be disease free and off treatment for > or = 3 years.
* Uncontrolled intercurrent illness including but not limited to: ongoing or active infection, systemic congestive heart failure Class III or IV by NYHA criteria, unstable angina pectoris, or cardiac arrhythmia, or in patients status post allogeneic transplantation with uncontrolled graft versus host disease (GVHD).
* Pre-existing neuropathy grade III or greater.
* Pregnant or nursing.
* Known hypersensitivity to brentuximab vedotin, bendamustine, or mannitol.
* Known Human Immunodeficiency Virus (HIV) positive, or hepatitis A, hepatitis B or hepatitis C; if hepatitis Bsurface antigen positive or Bcore antibody positive must have normal liver function tests and be willing and able to take anti-hepatitis medication such as lamivudine or equivalent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of brentuximab vedotin and bendamustine (phase 1) | Up to 1.5 years
  The highest dose that does not cause unacceptable side effects.
Dose limiting toxicities (DLT) of brentuximab vedotin and bendamustine (phase 1) | Up to 1.5 years
  A toxicity that prevents further administration of the agent at that dose level.
Overall Response Rate for the combination of brentuximab vedotin and bendamustine (phase 2) | Up to 3 years
  The percentage of subjects whose cancer shrinks or disappears after study treatment - Complete Response and Partial Response.

SECONDARY OUTCOMES:
Duration of Response (DoR) (phase 1) | Up to 3 years
  Time from documentation of tumor response to disease progression.
Progression free survival (PFS) (phase 1) | Up to 3 years
  The length of time during and after the study treatment that a subject lives with the disease but it does not get worse.
Overall Survival (OS) (phase 2) | Up to 3 years
  The length of time from either the date of diagnosis or the start of study treatment that subjects diagnosed with the disease are still alive.

OTHER OUTCOMES:
Serum Tarc levels | Up to 3 years
  This is designed to measure the response to study treatment if the level declines.
Level of peripheral blood lymphocyte expression of programmed death-1 (PD-1) | Up to 3 years
  The level will be evaluated as a function of response to therapy with brentuximab vedotin and bendamsutine.
Decline in serum levels of IL-10 and IL-6 | Up to 3 years
  The decline will be evaluated as a function of response to therapy with brentuximab vedotin and bendamsutine.

CONTACTS AND LOCATIONS:
Overall Officials: Owen A O'Connor, MD, Ph.D., Principal Investigator — Columbia University
Locations (3):
- Center for Lymphoid Malignancies at CUMC, New York, New York, United States
- Canada (2):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connor OA, Lue JK, Sawas A, Amengual JE, Deng C, Kalac M, Falchi L, Marchi E, Turenne I, Lichtenstein R, Rojas C, Francescone M, Schwartz L, Cheng B, Savage KJ, Villa D, Crump M, Prica A, Kukreti V, Cremers S, Connors JM, Kuruvilla J. Brentuximab vedotin plus bendamustine in relapsed or refractory Hodgkin's lymphoma: an international, multicentre, single-arm, phase 1-2 trial. Lancet Oncol. 2018 Feb;19(2):257-266. doi: 10.1016/S1470-2045(17)30912-9. Epub 2017 Dec 21. PMID 29276022